CLINICAL TRIAL: NCT07259187
Title: A Retrospective Analysis of Complications and Survival of Teeth Restored With Single Crowns Following Crown Lengthening
Brief Title: Retrospective Analysis of Complications and Survival of Teeth Restored Following Crown Lengthening
Status: Completed | Type: Observational
Sponsor: Mohammed Bin Rashid University of Medicine and Health Sciences (Other)
Responsible Party: Principal Investigator, Maanas Shah, Assistant Professor, Mohammed Bin Rashid University of Medicine and Health Sciences
Other Study IDs: MBRU-IRB-2022-97
Record Dates: First submitted 2025-11-19; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-10

CONDITIONS: Limited Tooth Structure; Crown Lengthening
Keywords: complications; survival rate; crown lengthening; endodontics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- single crowns post surgical crown lenghtening: Patients who underwent surgical crown lengthening prior to receiving single-crown restorations were contacted to participate in the study. The restored teeth were clinically and radiographically examined. Demographic data, patient- and tooth- related details, prevalence of prosthodontic, periodontal, and/or endodontic complications, as well as failure rate with underlying reason were documented and analyzed.
  Interventions: Diagnostic Test: Periapical radiograph

INTERVENTIONS:
Diagnostic Test: Periapical radiograph — Clinical and radiographic examinations were completed for the treated teeth. For participants who had radiographs within past one year of examination no further radiographs were obtained. Demographic parameters, systemic and patient-related factors such as smoking, diabetes mellitus, parafunctional habits (self-reported or diagnosed bruxism and clenching), location of tooth (maxilla or mandible, anterior or posterior), history of treated periodontitis, history of endodontic treatment, and history of regular dental attendance were documented. Furthermore, periodontal status was evaluated by assessing mobility, probing pocket depth, bleeding index, plaque index, restorative margin position in relation to the gingival margin, and crown to root ratio based on periapical radiographs taken using long-cone parallel technique. In addition, prosthetic factors including crown material and opposing dentition, namely tooth, crown, or removable partial denture were recorded.

SUMMARY:
The ultimate goal for every dental restoration is to restore and maintain the dentition's functionality along with preserving periodontal support. The long-term success of a restored tooth depends on the retention of a healthy periodontium. When restoring a short clinical crown, the clinician may contemplate placement of subgingival margin to gain additional length for retention purposes. Thus, crown lengthening procedure is performed to gain access to the natural tooth structure while maintaining the periodontal health and to increase the retention of the restoration. A full crown restoration is needed to protect the compromised tooth from fracture. The prognosis of these teeth depends on the long-term success rate of each component of the overall treatment and the follow up maintenance.

In order to assist dentists to make an evidence-based decision during treatment planning, this retrospective study aims to investigate the complications and survival rate of the teeth receiving crown following crown lengthening.

DETAILED DESCRIPTION:
The aim of this retrospective study was to evaluate the survival rates and complications of structurally compromised teeth restored with full-coverage crowns following crown lengthening procedure (CLP), in a postgraduate dental setting.

In this retrospective study the records of patients who received surgical CLP prior to receiving full coverage crowns at X hospital between January 2011 to January 2021 were obtained and reviewed by A.AH and F.AR for possible inclusion in the study. Retrospective data were collected manually from digital records of registered patients (Dental4windows, Centaur Software Development Co Pty Ltd., Australia). All personal information is de-identified and securely stored with a study code number. The data were then organized into categories based on a pre-determined form for single crowns with CLP .

The calculation of sample size was based on a 10-year survival rate of 78.4% tooth preservation after crown lengthening procedure and restorative treatment in department of periodontics and oral medicine at the school of dentistry of the university of Michigan (where p is the prevalence of crown after crown lengthening, d is the precision of the estimate, and z_(α/2)^2 is the quartile of the 95% confidence interval).

Using the above equation and data from the aforementioned study, the sample size needed is determined to be 260 teeth.

Statistical Analysis The collected data will be transferred to Statistical Package for Social Sciences (SPSS) for Windows (IBM- SPSS) version 25.0 (SPSS Inc., Chicago, IL, USA) for statistical analysis.

Significance for statistical analysis will be set at P < 0.05. Chi-square analysis will be used to measure the association strength between the frequency of both the survival of crown after crown lengthening and the complications. Kaplan-Meier will be used for analysis of the survival and Logistic regression will be used for the potential risk factors. P values <0.05 will be considered as a statistically significant.

ELIGIBILITY:
Inclusion Criteria: Patients were included in the study if they met all the following conditions:

* Setting and Providers: The tooth received crown lengthening surgery (CLP) performed by postgraduate residents in Periodontology and subsequent definitive crown placement by postgraduate residents in Prosthodontics at X Hospital.
* Patient Characteristics:

Age between 18 and 70 years at the time of the CLP. Able and willing to participate, with written informed consent obtained.

- Follow-up and Documentation Requirements: A minimum of 12 months had elapsed since placement of the definitive crown at the time of data collection. Baseline intraoral radiographs available prior to CLP to document periodontal and structural condition.

- Tooth-Level Clinical Criteria: Tooth mobility not exceeding Miller Class I at baseline. A planned or anticipated crown-root ratio ≥1:1 following CLP based on clinical and radiographic evaluation.

Exclusion Criteria: Patients were excluded if any of the following conditions applied:

* Procedure Purpose or Type: CLP performed exclusively for aesthetic indications.
* Cases involving intentional endodontic treatment and CLP performed solely to correct supra-eruption for prosthetic clearance (i.e., without biological indication).
* Baseline Dental and Periodontal Condition:

Teeth exhibiting furcation involvement at baseline. Mobility greater than Miller Class I preoperatively.

* Teeth functioning as abutments for fixed dental prostheses, due to altered biomechanical loading.
* Treatment Completion and Record Accuracy:

Absence or incompleteness of clinical or radiographic documentation prior to CLP. Incomplete endodontic, periodontal, or definitive restorative treatment at the time of review.

* The final restoration was not a full-coverage definitive crown.
* Follow-up and Participant Availability:

Follow-up duration less than 12 months after crown placement. Patients who declined participation or could not be contacted for consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were included if both the CLP and crown placement procedures were performed by postgraduate residents in periodontology and prosthodontics departments, respectively, at X hospital. All patients aged between 18 and 70 years at the time of treatment, and for whom at least one year had elapsed since definitive crown placement
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Teeth survival | 1 year or more postintervention
  tooth survival was defined as tooth remaining in situ with or without complications

CONTACTS AND LOCATIONS:
Overall Officials: Maanas Shah, BDS MSD CAGS MRACDS, Principal Investigator — Mohammed Bin Rashid University of Medicine and Health Sciences
Locations (1):
- Dubai Dental Hospital, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided
The authors have decided not to share individual participant data (IPD) because the dataset contains clinical information derived from patient records within an academic training setting, and complete anonymization cannot be fully guaranteed. In addition, institutional and ethical board policies restrict external sharing of patient-level data to protect participant confidentiality. Summary data supporting the findings of this study are available within the manuscript and supplementary materials.

REFERENCES:
- [Result] Ashnagar S, Barootchi S, Ravida A, Tattan M, Wang HL, Wang CW. Long-term survival of structurally compromised tooth preserved with crown lengthening procedure and restorative treatment: A pilot retrospective analysis. J Clin Periodontol. 2019 Jul;46(7):751-757. doi: 10.1111/jcpe.13124. Epub 2019 May 31. PMID 31050812